CLINICAL TRIAL: NCT00819871
Title: Association of NFKB1 -94 Polymorphism With Lung and/or Kidney Injury After Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Nuclear Factor Kappa-B (NFKB1) Polymorphism and Organ Injury After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jia-feng Wang, M.D., Changhai Hospital
Other Study IDs: PCSP-NFKB1
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Single Nucleotide Polymorphism; Acute Lung Injury; Kidney Injury
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3ml blood before surgery, after surgery and 24h after surgery respectively
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- PLI: patients with postoperative lung injury
- without PLI: patients without postoperative lung injury
- PLI/PKI: patients with at least one organ injury of lung or kidney after surgery
- without PLI/PKI: patients without lung or kidney injury after surgery

SUMMARY:
NFKB1 -94ins/del polymorphism has been reported to be associated with reduced promoter activity of NFKB1 and several clinical diseases, but the clinical results cannot always be replicated. Besides, mutate allele is associated with alleviated inflammation in ulcerative colitis and some tumors, but aggravated inflammation in ARDS. The clinical value of this polymorphism remains controversial. This study was performed to investigate the association of NFKB1 -94ins/delATTG polymorphism with lung and/or kidney injury after cardiac surgery with CPB.

ELIGIBILITY:
Inclusion Criteria:

* Chinese Han unrelated population
* undergoing elective cardiac surgery with CPB

Exclusion Criteria:

* malignant tumor
* autoimmune disease, immunodeficiency or immunosuppressive therapy
* chronic renal disease (glomerular filtration rate < 60ml/(min•1.73m2)) or liver dysfunction (Child Pugh classification>A)
* COPD, tuberculosis or other chronic pulmonary diseases
* anemia with hemoglobin lower than 90mmHg
* bleeding disorders
* postoperative pericardial tamponade requiring re-operation
* postoperative low cardiac output syndrome or acute pulmonary edema after left cardiac failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese Han patients undergoing elective cardiac surgery with CPB
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
lung injury and/or kidney injury after cardiac surgery with cardiopulmonary bypass | 24h after cardiac surgery

SECONDARY OUTCOMES:
circulating level of CRP, TNF-alpha, IL-10; APACHE Ⅱ score; duration of ICU stay and hospitalization; death in 28 days | one month after cardiac surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

REFERENCES:
- [Result] Wang JF, Bian JJ, Wan XJ, Zhu KM, Sun ZZ, Lu AD. NFKB1-94ins/del polymorphism is not associated with lung injury after cardiopulmonary bypass. Anaesthesia. 2010 Feb;65(2):158-62. doi: 10.1111/j.1365-2044.2009.06186.x. Epub 2009 Nov 25. PMID 19995347